CLINICAL TRIAL: NCT02764346
Title: iCanCope With Pain: Usability and Feasibility Testing of a Smartphone Application to Manage Pain in Youth With Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Alberta Children's Hospital (Other); British Columbia Children's Hospital (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Clinician Scientist, Clinical Nurse Specialist/NP, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000049274
Record Dates: First submitted 2016-04-27; First posted 2016-05-06 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Arthritis; Self-management; Pain
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- iCanCope app (Experimental): iCanCope app
  Interventions: Behavioral: iCanCope app
- Attention control app (Active Comparator): Control group: iCanCope attention control app
  Interventions: Behavioral: iCanCope attention control app

INTERVENTIONS:
Behavioral: iCanCope app — In addition to standard medical care, adolescents in the experimental group will receive access to the "iCanCope" smartphone app for 8 weeks. The app consists of daily pain symptom tracking (pain intensity, sleep, mood, physical activity, and fatigue), goal setting, in-the moment coping strategies, as well as a social community component.
  Arms: iCanCope app
Behavioral: iCanCope attention control app — The control group is designed to control for the potential effects on outcomes of time, attention, and smartphone use during the intervention. In addition to standard medical care, adolescents in the attention control group will receive access to the "iCanCope" control app, with limited functionality.
  Arms: Attention control app

SUMMARY:
This study will look at the use and impact of smartphone application (app) for adolescents with ongoing pain caused by their juvenile idiopathic arthritis (JIA).The current project will include three studies. First, the investigators conducted usability sessions with adolescents with JIA to refine the app so that it is usable, acceptable and understandable. The aim of this study is to look at (a) how regularly the "iCanCope with Pain" app is used and (b) any effect the app has on young people's health. This study will compare two groups of young people: one that is using the new app, and one that receives usual medical care.

ELIGIBILITY:
Inclusion Criteria

1. Aged 12-18 years
2. Diagnosed with JIA (36) as per their rheumatologist
3. Able to speak and read English
4. Have self-reported average arthritis-related pain in the past week of >3 on 10cm visual analogue scale (VAS)
5. Willing to complete online study outcome measures

Exclusion Criteria:

1. Moderate to severe cognitive impairments as per their healthcare provider
2. Major co-morbid psychiatric [conversion disorder, depression, anxiety disorder] illnesses that may impact their ability to understand and use the "iCanCope with Pain" intervention as per their rheumatologist
3. Received more than 4 CBT sessions for pain management in the past 6 months, as per their healthcare provider and self-report
4. Patients from the department of haematology/oncology

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Participant accrual rate | 8 weeks
  Centrally tracked by the clinical research project coordinator
Number of issues or difficulties in implementing the intervention | 8 weeks
  The intervention fidelity log will track any issues or difficulties encountered during implementation of the intervention, control strategy, or outcome measures will be tracked throughout the study by the CRPC.
Acceptability of intervention | 8 weeks
  Participants in the intervention arm will complete the Acceptability e-scale (AES) post-intervention. In addition, a subset of participants from the intervention group will be offered to participate in a qualitative feedback interview to further explore acceptability of the intervention.
Frequency of login per user | 8 weeks
  Measured through the iCanCope server.
Adherence | 8 weeks
  Adherence will be determined using Google Analytics.
Adverse Events | 8 weeks
  Adverse events will be tracked using an adverse event form
Participant dropout rate | 8 weeks
  Centrally tracked by clinical research project coordinator
Satisfaction of intervention | 8 weeks
  A subset of participants from the intervention group will be offered to participate in a qualitative feedback interview to further explore satisfaction of the intervention.

SECONDARY OUTCOMES:
Pain | 8 weeks
  Pain will be measured using the Standardized Universal Pain Evaluations for Rheumatology providers for children and youth (SUPERKIDZ). It consists of 4 domains: pain intensity and location (5 items), fatigue (1 item), pain interference/evaluative dimension (10 items), and affective/emotional dimension (4 items) for children > 8 years. This online measure takes 3 - 5 minutes to complete, and has evidence of test-retest reliability, construct validity, and responsiveness.
Pain-Related Activity Limitations | 8 weeks
  Pain-related activity limitations will be measured using the Child Activity Limitations Interview (CALI-21). This is a well-validated 21-item self-report scale divided into (i) active (e.g., gym, sports) and (ii) routine (e.g., schoolwork, reading) activity subscales.
Pain coping | 8 weeks
  Pain coping will be measured using the Pain Coping Questionnaire which is an internationally used measure of pain coping strategies in pediatric populations. Respondents indicate on a 5-point scale how often they use a given type of coping strategy from among 8 different categories. Three higher order factor-derived subscale scores will be used for analyses, including approach coping (e.g., problem-solving), problem-focused avoidance coping (e.g., cognitive distraction), and emotion-focused avoidance coping (e.g., catastrophizing). The measure is considered to meet psychometric criteria for a "well-established" coping measure and is responsive to pain coping interventions.
Health-Related Quality of Life (HRQoL) | 8 weeks
  HRQoL will be measured using the PedsQL 3.0 Arthritis Module, which measures the potential impact on quality of life of having arthritis in childhood. The scale has 22 items and evaluates the severity of perceived problems with disease symptoms, daily activity limitations, treatments, worry/anxiety, and communication.
Health care utilization form | 8 weeks
  This will be used to measure direct health care costs and patient/family out of pocket costs related to arthritis care
Health Utility Index | 8 weeks
  Used to calculate quality adjusted life years (QALYs)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lalloo C, Harris LR, Hundert AS, Berard R, Cafazzo J, Connelly M, Feldman BM, Houghton K, Huber A, Laxer RM, Luca N, Schmeling H, Spiegel L, Tucker LB, Pham Q, Davies-Chalmers CC, Stinson JN. The iCanCope pain self-management application for adolescents with juvenile idiopathic arthritis: a pilot randomized controlled trial. Rheumatology (Oxford). 2021 Jan 5;60(1):196-206. doi: 10.1093/rheumatology/keaa178. PMID 32613229